CLINICAL TRIAL: NCT00673400
Title: Morbidity and Functional Outcome of Stapled TransAnal Rectal Resection (STARR) With Contour® TranstarTM in Obstructed Defecation
Brief Title: Stapled TransAnal Rectal Resection (STARR) With Contour® TranstarTM
Acronym: STARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, F. Hetzer, Leitender Arzt, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARR
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Obstructed Defecation Syndrome; Rectocele; Intussusception; SNS
Keywords: Obstructed defecation syndrome; ODS; Rectocele; Intussusception; STARR
MeSH Terms: conditions — Rectocele; Intussusception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stapled transanal rectum resection (Other): patients operated with stapled transanal rectum resection
  Interventions: Procedure: Stapled transanal rectum resection

INTERVENTIONS:
Procedure: Stapled transanal rectum resection — Contour Transtar-STR5G (Ethicon EndoSurgery Inc., Cincinnati, OH).The circular anal dilator is fixed to perianal skin.Rectal intussusception is evidenced with a swab.The first stitch is placed superficial on top of the intussusception. The procedure is performed 5to6 times counterclockwise.A final stitch for first radial cut at 3 o'clock.The device is introduced into the rectum. This cut opens the prolapse. Check with a finger the vagina. The device is then closed and fired. After replacing the cartridge, the device is introduced in the rectum, placed parallel to the circular anal dilator and moved counter clockwise with 4to6firings to complete the resection. Additional stitches across the staple line to assure haemostasis.

SUMMARY:
The stapled transanal rectal resection (STARR procedure) is an effective treatment for obstructed defecation syndrome (ODS) caused by intussusception and rectocele. Recently a new technique has been developed using the new Contour® TranstarTM stapler, which was specifically designed to facilitate the STARR procedure. The investigators would like to evaluate the morbidity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Rectocele
* Intussusception

Exclusion Criteria:

* Non operability
* inflammatory bowel disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franc Hetzer, MD, Principal Investigator — Cantonal Hospital St. Gallen, Department of Surgery
Locations (1):
- Department of Surgery, Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Wolff K, Marti L, Beutner U, Steffen T, Lange J, Hetzer FH. Functional outcome and quality of life after stapled transanal rectal resection for obstructed defecation syndrome. Dis Colon Rectum. 2010 Jun;53(6):881-8. doi: 10.1007/DCR.0b013e3181cdb445. PMID 20485001

RESULTS

PARTICIPANT FLOW:
Groups:
- Stapled TransAnal Rectal Resection: patients were operated by stapled transanal rectal resection
Period: Overall Study
Arm/Group | Stapled TransAnal Rectal Resection
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stapled TransAnal Rectal Resection
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 52

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life
Description: Quality of life is measured by Fecal incontinence quality of life (FIQL)
  Possible range of score 0 - 4 (Depression/Self perception 4.4)
  0 = worst condition
  * Fecal Incontinence Quality of Life (FIQL) (Rockwood, Dis Colon Rectum (2000) 43:9)
Time Frame: 6 months after intervention
Population: Participating in the FIQL survey was voluntarily. Some patients did not participate at all, some did not answer all questions. Patients answering >=50% of questions of a domain were counted as participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Before Surgery; 6 Months After Surgery: outcome measured within one month before surgery
Arm/Group | Before Surgery | 6 Months After Surgery
Number analyzed (Participants) | 35 | 41
units on a scale
  Lifestyle (LS) | 3.2 [2.4 to 3.6] | 3.7 [2.4 to 4.0]
  Coping/behavior (C/P) | 2.8 [2.1 to 3.6] | 3.3 [2.2 to 4.0]
  Depression/self-perception (D/S) | 3.3 [2.3 to 3.9] | 3.9 [3.1 to 4.1]
  Embarrassment (E) | 3.3 [2.3 to 4.0] | 4.0 [3.7 to 4.0]
Statistical Analysis 1: Comparison: Before Surgery vs 6 Months After Surgery; Lifestyle (LS); Test type: Superiority or Other; p = 0.1340, Wilcoxon (Mann-Whitney) — based on 28 pairwise matches; matched pair test, two-sided, exact method
Statistical Analysis 2: Comparison: Before Surgery vs 6 Months After Surgery; Coping/behavior (C/B); Test type: Superiority or Other; p = 0.088, Wilcoxon (Mann-Whitney) — based on 29 matched pairs; matched pair test, two-sided, exact method
Statistical Analysis 3: Comparison: Before Surgery vs 6 Months After Surgery; Depression/self-perception (D/S); Test type: Superiority or Other; p = 0.0012, Wilcoxon (Mann-Whitney) — based on 30 matched pairs; matched pair test, two-sided, exact method
Statistical Analysis 4: Comparison: Before Surgery vs 6 Months After Surgery; Embarrassment (E); Test type: Superiority or Other; p = 0.0074, Wilcoxon (Mann-Whitney) — based on 30 matched pairs; matched pair test, two-sided, exact method

2. Secondary Outcome: Morbidity
Description: Surgical complications after treatment according to Dindo (Ann Surg (2004) 240:205)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Stapled TransAnal Rectal Resection
Number analyzed (Participants) | 52
participants
  overall | 6
  Urinay retention (Dindo IIIa) (within 30 days) | 1
  self limiting rectal bleeding (Dindo I)(6 weeks) | 2
  Pain from residual staple (Dindo IIIa)(6 weeks) | 2
  Perianal venous thrombosis (Dindo IIIa) (5 weeks) | 1

3. Secondary Outcome: Hospitalization
Description: Length of hospital stay (Date of release - Date of admission + 1)
Time Frame: 1 day to 1 year (until release from hospital)
Measure: Median (Full Range); unit: days
Arm/Group | Stapled TransAnal Rectal Resection
Number analyzed (Participants) | 52
days | 5 [2 to 29]

4. Other Pre Specified Outcome: Severity of Symptoms Score
Description: Score based on the severity of 9 symptoms of bowel movement (physician administered)
  (0 - 36, no symptoms = 0)
  Dis Colon Rectum 39:681 (DOI: 10.1007/BF02056950)
Time Frame: before surgery - 6 weeks - 3 months - 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- 6 Weeks After Surgery: outcome measured 6 weeks after surgery
- 3 Months After Surgery: outcome measured 3 months after surgery
- 6 Months After Surgery: outcome measured 6 months after surgery
Arm/Group | Before Surgery | 6 Weeks After Surgery | 3 Months After Surgery | 6 Months After Surgery
Number analyzed (Participants) | 52 | 52 | 46 | 25
units on a scale | 15 [13 to 17] | 4 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Before Surgery vs 6 Weeks After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method
Statistical Analysis 2: Comparison: Before Surgery vs 3 Months After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method
Statistical Analysis 3: Comparison: Before Surgery vs 6 Months After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method

5. Other Pre Specified Outcome: Obstructive Defecation Syndrome Score
Description: Score based on severity or frequency of 9 symptoms of obstructive defecation (physician administered)
  (0 - 40, no symptoms = 0)
  Dis Colon Rectum 51:348(DOI: 10.1007/s10350-007-9115-1)
Time Frame: before surgery - 6 weeks -3 months - 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Before Surgery | 6 Weeks After Surgery | 3 Months After Surgery | 6 Months After Surgery
Number analyzed (Participants) | 52 | 52 | 46 | 25
units on a scale | 16 [14 to 18] | 5 [3 to 6] | 4 [3 to 5] | 5 [2 to 7]
Statistical Analysis 1: Comparison: Before Surgery vs 6 Weeks After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method
Statistical Analysis 2: Comparison: Before Surgery vs 3 Months After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method
Statistical Analysis 3: Comparison: Before Surgery vs 6 Months After Surgery; Test type: Superiority or Other; p < 0.0000001, Wilcoxon (Mann-Whitney); two-sided, paired test, exact method

6. Other Pre Specified Outcome: SF36 Component Summary Scores
Description: Quality of life short form 36 version 2(SF36v2) standard form
  PCS: physical component summary score (range 1 to 81, with 81 being the best) MCS: mental component summary score (range -9 to 82, with 82 being the best)
  A score of 50 correlates with the result of a healthy standard US population (score transformation to a mean of 50 and a standard deviation of 10)
  Ware JE, Kosinski M, Dewey JE. How to Score Version 2 of the SF-36® Health Survey. Lincoln, RI: QualityMetric Incorporated, 2000.
Time Frame: Before surgery - 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Before Surgery | 6 Months After Surgery
Number analyzed (Participants) | 35 | 41
units on a scale
  Physical component summary (PCS) | 51 [43 to 55] | 52 [35 to 55]
  Mental component summary (MCS) | 39 [33 to 51] | 53 [40 to 58]
Statistical Analysis 1: Comparison: Before Surgery vs 6 Months After Surgery; Physical component summary (PCS); Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney) — based on 28 pairwise matches; matched pair test, two-sided, exact method
Statistical Analysis 2: Comparison: Before Surgery vs 6 Months After Surgery; Mental component summary (MCS); Test type: Superiority or Other; p = 0.010, Wilcoxon (Mann-Whitney) — based on 28 pairwise matches; matched pair test, two-sided, exact method

ADVERSE EVENTS:
Time Frame: 1 year
Description: Grading of adverse events according to Accordion/Dindo Scale see also secondary outcome: morbidity (Ann Surg (2004) 240:205)
Arm/Group | Stapled TransAnal Rectal Resection
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 4/52
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stapled TransAnal Rectal Resection (N=52)
persisting pain due to residual staples (Injury, poisoning and procedural complications) | 2 (2) — Dindo grade IIIa: intervention without general anesthesia
thrombosis (Blood and lymphatic system disorders) | 1 (1) — perianal venous thrombosis 5 weeks postoperatively Dindo grade IIIb: incision under general anesthesia
urinary retention (Renal and urinary disorders) | 1 (1) — Dindo grade IIIa: intervention without general anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes